CLINICAL TRIAL: NCT06367790
Title: Plyometry and Tapping in the Functional Improvement of Non-professional Basketball Players. Randomised Clinical Study
Brief Title: Plyometry and Tapping in the Functional Improvement of Non-professional Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Bask-Pliomet
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-04

CONDITIONS: Basketball Players
Keywords: Basketball; Plyometric exercises; Dry needling; Range of motion; Vertical jump.
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention period will last 4 weeks, with a periodicity of 2 weekly sessions of 30 minutes each. All interventions will take place in the sports facilities of both clubs. The interventions will be carried out by the principal investigator of the study. The 10 players assigned to the experimental group will perform plyometric exercises and will undergo dry needling of the gastrocnemius (gastrocnemius muscle) and the control group (plyometric exercises and dry needling of the gastrocnemius muscle).
  Interventions: Other: Experimental group
- Control group (Active Comparator): The 10 players assigned to the control group will perform plyometric exercises.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Experimental group — The athletes included in the experimental group will undergo an intervention using a plyometric exercise protocol, 2 days a week, and dry needling of the gastrocnemius muscles will be applied in a weekly session.
  To perform the dry needling intervention, 0.3x50mm disposable steel needles will be used, applying the "quick in-and-out" technique. To do this, first of all, the intervention area will be cleaned with alcohol and sterile gloves will be used to perform the manoeuvre in complete safety. The active or latent trigger point is then located within the taut band by inserting the needle deeper and deeper, and then moving the needle up and down in search of a local contraction response. A maximum of 8 insertions or up to the athlete's tolerance limit will be applied.
  Arms: Experimental group
Other: Control group — The athletes included in the control group will perform an intervention using a plyometric exercise protocol, 2 days a week, under the same conditions as the experimental group.
  Arms: Control group

SUMMARY:
Introduction. In basketball, the lower extremities have the highest prevalence of injury, regardless of gender and professional category.

Objective. To analyse the efficacy of a physiotherapy intervention using a protocol of plyometric exercises and dry needling in non-professional basketball athletes.

Methods. Randomised clinical study. 20 players will be randomised to an experimental group (plyometric exercises and dry needling of the gastrocnemius muscles) and a control group (plyometric exercises). The intervention will include 8 sessions over 4 weeks. The study variables will be: range of motion in dorsal flexion in loading (Leg Motion®) and unloading (goniometer) and vertical jump (MyJump2®).

Expected results. An intervention of plyometric exercises and dry needling produces significant differences in range of motion and vertical jump in basketball players, compared to the isolated administration of plyometric exercises.

ELIGIBILITY:
Inclusion Criteria:

* Non-professional basketball players who are in competition.
* Subjects over 18 years of age
* Athletes competing in the first men's division of the basketball federation of the Region of Murcia.
* Sign the informed consent document.

Exclusion Criteria:

* Subjects who are injured at the time of data collection.
* Subjects who are unable to attend all training sessions during the duration of the research.
* Athletes with apprehension to dry needling.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline range of motion in loaded dorsal flexion after treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  Loaded dorsiflexion of the ankle will be assessed using the Leg Motion® device. This test consists of placing the athlete barefoot with the foot on the measuring scale of the instrument, requesting maximum knee flexion without lifting the heel. The test is performed 3 times and the average value is used in the data analysis. The unit of measurement is the maximum distance, measured in centimetres, between the toe and the metal bar. The greater the distance, the greater the dorsiflexion in ankle loading.

SECONDARY OUTCOMES:
Change from baseline range of motion in unloaded dorsal flexion after treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  Passive dorsiflexion of the ankle shall be measured in the supine position using a universal goniometer. For this assessment, the axis of the goniometer is placed over the centre of the lateral malleolus, while the fixed arm is placed parallel to the fibula towards the head of the fibula, and the movable arm is placed parallel to the 5th metatarsal. The unit of measurement is a value in degrees, where the higher the graduation, the greater the ankle dorsiflexion.
Change from baseline vertical jump after treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up visit
  The variable vertical jump height will be measured with the MyJump2® application. In this test, the evaluator stands 1.5 metres away from the athlete with the mobile phone at ground level. The player must perform a jump with both feet on the ground and the hands on the hips. When the athlete is in the flight phase, he/she should have both legs extended, while when landing, the first contact should be with the metatarsals. The unit of measurement of this tool is in centimetres, where the greater the distance, the greater the vertical jump.

CONTACTS AND LOCATIONS:
Locations (1):
- Rubén Cuesta-Barriuso, Oviedo, Principality of Asturias, Spain